CLINICAL TRIAL: NCT02953080
Title: Improving Outcomes in HIV Patients Using Mobile Phone Based Interactive Software Support
Acronym: Callforlife
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ST/163/2016
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-01

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — CD56 Antigen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Call for Life Mobile phone support (Active Comparator): The intervention is "Call for life mHealth adherence support tool " through basic mobile phone-based interactive voice response.
  Interventions: Other: Call for life mHealth adherence support
- Standard of Care (No Intervention): No call for life Uganda: Patients are randomized to standard of Care

INTERVENTIONS:
Other: Call for life mHealth adherence support — Daily/ weekly pill reminder support Health Info-tips Appointment visit reminders Self-reported symptom support
  Other Names: mHealth system
  Arms: Call for Life Mobile phone support

SUMMARY:
Current estimates point towards a huge increase in the number of people that are eligible to start ART in Uganda and globally. As many of the newly eligible patients are largely asymptomatic, there are concerns about adherence and retention of these individuals and especially those starting ART with a higher CD4 counts. Urgent information is required to plan for implementation of most recent WHO and National guidelines in the most cost effective manner as well as maximizing retention of HIV positive individuals in care and achieving virological suppression.

The investigators plan to undertake research designed to see if investigators can optimize adherence, virological outcomes and HIV knowledge, in order to give an overall increased quality of life in vulnerable populations starting or established on ART in Kampala, Uganda. The investigators will test implementation of an open source software-based tool to send text messages and to give access to an interactive voice response system using patients' mobile phones.

The investigators' aim to undertake an open labelled randomised trial at two sites: the IDI which is an urban centre of excellence in HIV care, and Kasangati Health Centre, which is a peri-urban public health care facility. The project aims to enrol HIV positive patients starting ART, already established on first line ART or switching to second line ART, including special populations (pregnant women, discordant couples and young people). The estimated length of the project is 30 months. The technology to be evaluated in this study is based on CONNECT FOR LIFETM m-health technology (CFL2015.01 or higher), which provides text messages or Interactive Voice Response (IVR) functionalities, and allows a computer to interact with humans through the use of voice and tones input via keypad and offers pill reminders, clinic visit reminders, health tips and support symptom reporting.

Primary Objective is to determine the effect of the CFL2015.01 tool on quality of life of HIV patients receiving care at IDI and Kasangati HCIV. At the start of the intervention, all patients will undergo quality of life assessment, which will be repeated at months 6, 12, 18 and 24 months. The scores will be compared to assess the effect of the tool on quality of life. The Secondary Objectives are virological outcomes baseline, 6, 12,18 and 24 months, retention in care, aversion of early treatment failure, disease knowledge, clinic attendance and cost analysis.

DETAILED DESCRIPTION:
CALL FOR LIFE UGANDATM Janssen Global Public Health Research and Development, in close collaboration with the Infectious Disease Institute Kampala (IDI), has developed Call for Life Uganda tailored to the needs of PLHIV in Uganda. Call for Life UgandaTM is based on the CONNECT FOR LIFETM technology (CFL2015.01 or higher version) and the MOTECH platform, an open source platform developed by Grameen Foundation and the University of Southern Maine with financial support from the Bill and Melinda Gates Foundation, and was released under the terms of the MOTECH open source license agreement.

All patients consenting will; At enrolment receive detailed information from a nurse/counsellor on the Call for Life UgandaTM system and how it operates Receive calls or text messages from Call for Life UgandaTM will include recording of self-reported adherence (soliciting active feedback via keypad) and symptom management triggering alerts for the clinic.

STUDY PROCEDURES Screening The subjects will be screened and enrolled over a period of 6 months These are the screening procedures oAll consecutive eligible patients will be approached for participation in the study.

oFor patients interested in participating the inclusion and exclusion criteria will be ascertained.

oThe patients will receive information about the study by the study nurse or counselor Patients who agree to participate in the study will sign the informed Follow-up Visit The participants will come to the clinic monthly or 2 monthly to pick up their ART and concomitant medications (non-study visits).

The participants will come for their study follow up visits every 6 months Every 6 months The patients will be assessed by the study staff.

* The study doctor will collect General Medical History and perform Physical Examination and enter it in an electronic CRF.
* The counsellor will collect the Quality of life and Knowledge questionnaires and enter them in an electronic CRF.

At baseline, 6, 12,18 and 24 months the following samples will be collected;

* Viral load
* Storage plasma (1 aliquot) serum (3 aliquots)

Additional procedures Resistance testing: It will be done on stored samples

* Baseline Resistance testing will be carried out if subsequent viral failure in order to investigate transmitted resistant virus
* Biological samples will also be stored at 6, 12,18 and 24 months and resistance testing carried out in case of viral load >1,000 copies/ml

Subject Withdrawal Subjects may withdraw from the study at any time at their own request, or they may be withdrawn at any time at the discretion of the investigator for safety or behavioral reasons, or the inability of the subject to comply with the protocol required schedule of study visits or procedures.

SAFETY ASSESSMENT Safety monitoring for this study will focus on unanticipated problems involving risks to participants, including unanticipated problems that meet the definition of a serious adverse event.

DATA ANALYSIS/STATISTICAL METHODS Based on a pre and post ART assessment in Burkino Faso and Uganda, it is anticipated that the quality of life score (MOS-HIV) in ART naïve patients will increase at least by 15 points for physical health summary (PHS) between baseline and 12 months ART use. We estimate there will be an additional 5 points improvement in those receiving C4LTM which would give 20-point improvement for those on C4LTM and 15 points for those not on call for Life. In those already on ART, investigators estimate an improvement for those established on ART with a 5-point improvement for those on C4LTM and nil for those not accessing C4LTM. We also estimate a 5-point increase in mental health score in those receiving C4LTM compared to no change in those without C4LTM starting ART, and a lower improvement of 2 points in mental health score in those already on ART. The study is powered on the PHS for QOL. For a power of 0.9 and precision of 0.05 we would need a minimum of 273 in each arm (overall 546) patients, if the mean PHS among patients with C4L was 58.2 compared to 55.2 among patients without C4L. The investigators will include a 10% LTFUP/mortality rate to give a sample size of 600.

The composition of the study participants is estimated as 300 patients at Kasangati and 300 patients at IDI. With the proposed sample size, the numbers above depict over 90% power to test even the smallest differences in mean PHS at 12 months in the group of patients with and without C4L. The investigators also anticipate that it is possible to detect changes in MHS QOL with this sample Analysis of Primary Endpoint Scales to measure quality of life For this study we have chosen to use the Medical Outcomes Study (MOS-HIV) Health Survey which is the most widely used health related HRQoL measure in PLHIV.

The MOS-HIV scale was chosen because it has been validated in various settings including Uganda, has a Luganda language version, and was found to be useful in assessing HRQoL in PLHIV.

The MOS-HIV measures HRQoL in 11 areas: health perceptions, bodily pain, physical function, role function, social function, mental function, vitality, health distress, cognitive function, QoL, and health transition. One scores scale in a range from 0-100 with a higher score implying better health (41). In addition to these subscales, a Physical Health Summary score (PHS) and Mental Health Summary score (MHS) can be calculated.

Intra patient in QoL scores will be compared using Paired T-tests and overall change will be investigated. The effect of calendar time on QoL life scores will be accounted for during analysis. Furthermore, the changes and or effect of the intervention on different sub-groups of HIV positives patients will be carried. The effect of the intervention will also be compared between IDI and Kasangati sites. All analysis will be conducted using STATA, USA.

* Investigators will assess perceptions and attitudes to the Call for Life UgandaTM tool thorough focus group discussions and Key informant interviews, targeting each special population. We will use purposeful sampling and will continue until no new themes emerge. We will use NVIVO software for coding of themes.
* Cost analysis along with the study evaluation; appropriate and detailed cost evaluation will also be performed. It is anticipated that if the intervention is proved effective, a cost effective analysis would contribute to developing a sustainable scale up strategy for similar service across Uganda.

RADOMISATION Patients will randomly be assigned to either one of the two arms, that is, with and without CFL. To ensure that all patients in each of the arms are represented and equally balanced out in both arms, the study will use stratified randomization where each of the categories of patients at the start of the study will form the strata on interest. Within each stratum, the patients will be randomly assigned to C4L or no C4L. Randomization lists will be generated by an independent statistician and kept under lock and key in the two sites.

DATA PRIVACY Any and all data generated in IDI's use of Call for Life UgandaTM shall be owned solely by IDI. Therefore, IDI will take all reasonable steps to restrict disclosure of personal data including patient-identifiable to third parties.

In addition, the following Security Measures are in place to protect Patient's privacy when using Call for Life UgandaTM

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

  1. Evidence of a personally signed and dated informed consent document indicating that the subject (or a legal representative) has been informed of all pertinent aspects of the study.
  2. Patients who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
  3. Patients having the ability to use basic cell phone functions (e.g., being able to make and receive phone calls).
  4. Patients with access to a mobile phone (need to be able to answer the phone at a predetermined time slot and to be able to call the clinic if they are sick)
  5. Patients who are able to understand Luganda or Runyankole or English (as these are the languages of the overwhelming majority of patients at IDI and Kasangati and so will be used for the trial. If any other language has more than 30 patients who require it, the tool will be adapted to include this new language before the roll out of the tool to the entire clinic population

Exclusion Criteria:

1. Patient whose clinical condition interferes with appropriate use of cell phone (e.g., deafness, severe cognitive impairment)
2. Patients < 15 years unless emancipated minors as defined by Ugandan National Research Ethics Committee guidelines.
3. Patients who are enrolled in an interventional study at IDI
4. Patients who are not receiving standard first and second line treatment
5. Patients who are critically ill.

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2016-08-23 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Determine effect of Call for Life tool on physical quality of life of HIV patients receiving care at the 2 study sites | Month 06, Month 12, 18 and 24 MONTHS
  Change in physical health score by 5-point in those accessing Call for Life Uganda between baseline, 6 , 12, 18 and 24 months of Call for Life Uganda use, and comparison to those with no access to Call for Life UgandaTM at 6 and 12 months

SECONDARY OUTCOMES:
Determine effect of Call for Life tool on mental quality of life of HIV patients receiving care at the 2 study sites | Month 06, Month 12 , 18 and month 24
  Change in mental health score by 5-point in those accessing Call for Life Uganda between baseline, 18 and 24 months of Call for Life Uganda use, and comparison to those with no access to Call for Life UgandaTM at 18 and 24 months 2. Proportion of patients with viral load > 50 copies/ml at 18, and 24 months among patients using the Call for Life UgandaTM tool compared to those with no access to Call for Life UgandaTM
Determine effect of Call for Life tool on virological outcome and aversion of early treatment failure | Baseline, Month 6, 12, 18 and 24
  Viral load measurement at 6,12,18 and 24 months
Determine effect of Call for life Uganda, on retention in care at the 2 sites | 24 months
  Proportions of HIV patients retained in chronic care at the 2 sites
Determine effect of Call for life Uganda on attendance on scheduled appointment days +/- 2 working days | Month 06, 12, 18 and 24
  Clinic appointment keeping

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind Parkes-Ratanshi, Principal Investigator — Makerere University
Locations (1):
- Infectious Diseases Institute,Makerere University College of Health Sciences, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kajubi P, Parkes-Ratanshi R, Twimukye A, Bwanika Naggirinya A, Nabaggala MS, Kiragga A, Castelnuovo B, King R. Perceptions and Attitudes Toward an Interactive Voice Response Tool (Call for Life Uganda) Providing Adherence Support and Health Information to HIV-Positive Ugandans: Qualitative Study. JMIR Form Res. 2022 Dec 6;6(12):e36829. doi: 10.2196/36829. PMID 36472904
- [Derived] Naggirinya AB, Kyomugisha EL, Nabaggala MS, Nasasira B, Akirana J, Oseku E, Kiragga A, Castelnuovo B, King RL, Katabira E, Byonanebye DM, Lamorde M, Parkes-Ratanshi R. Willingness to pay for an mHealth anti-retroviral therapy adherence and information tool: Transitioning to sustainability, Call for life randomised study experience in Uganda. BMC Med Inform Decis Mak. 2022 Feb 26;22(1):52. doi: 10.1186/s12911-022-01782-0. PMID 35219309
- [Derived] Twimukye A, Bwanika Naggirinya A, Parkes-Ratanshi R, Kasirye R, Kiragga A, Castelnuovo B, Wasswa J, Nabaggala MS, Katabira E, Lamorde M, King RL. Acceptability of a Mobile Phone Support Tool (Call for Life Uganda) for Promoting Adherence to Antiretroviral Therapy Among Young Adults in a Randomized Controlled Trial: Exploratory Qualitative Study. JMIR Mhealth Uhealth. 2021 Jun 14;9(6):e17418. doi: 10.2196/17418. PMID 34121665
- [Derived] Byonanebye DM, Nabaggala MS, Naggirinya AB, Lamorde M, Oseku E, King R, Owarwo N, Laker E, Orama R, Castelnuovo B, Kiragga A, Parkes-Ratanshi R. An Interactive Voice Response Software to Improve the Quality of Life of People Living With HIV in Uganda: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Feb 11;9(2):e22229. doi: 10.2196/22229. PMID 33570497